CLINICAL TRIAL: NCT03822611
Title: Research on the Impact of Targeted Subsidies Within Open Defecation Free (ODF) Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Aquaya Institute (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Tetratech (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: WASHPaLS Subsidy Study
Record Dates: First submitted 2019-01-25; First posted 2019-01-30 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Sanitation

STUDY DESIGN:
Intervention Model Description: cluster Randomized controlled trial (c-RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted Subsidy (Experimental): In these communities, households identified as vulnerable receive a voucher for a free latrine sub-structure (slab + pit lining), redeemable with local sanitation suppliers.
  Interventions: Behavioral: Targeted Subsidy
- No subsidy (No Intervention): In these communities, no household receives a voucher.

INTERVENTIONS:
Behavioral: Targeted Subsidy — Voucher
  Arms: Targeted Subsidy

SUMMARY:
This study evaluates targeted subsidies as a strategy to improve sanitation infrastructure and behaviours in communities that have reached Open Defecation Free (ODF) status after a Community-Led Total Sanitation (CLTS) program. The investigator's hypothesis is that sanitation subsidies targeted at the most vulnerable households within ODF communities will increase and help sustain latrine coverage, quality, and use amongst the targeted households, and through a spill-over effect, amongst the rest of the community. Half of participating communities will receive the targeted subsidy, while the other half will not receive any treatment.

DETAILED DESCRIPTION:
Community-Led Total Sanitation (CLTS) is a widely used approach to eradicate open defecation in rural communities in developing countries. Using emotional triggers, CLTS promotes community self-help to build household latrines. In Ghana, where CLTS is part of the government's official sanitation strategy, a community is declared "Open Defecation Free" (ODF) when 80 percent of households own a latrine.

There is however evidence that open defecation persists in so-called "ODF" communities, especially as the most vulnerable households (the poorest of the poor) cannot afford to construct or maintain durable latrines. As a result, subsidies for these vulnerable households have been proposed as a strategy to promote the construction of durable latrines and help sustain safe sanitation behaviours in communities having received CLTS.

ELIGIBILITY:
This study is a cluster randomized controlled trial that will enroll entire communities. Within a community, only specific households will be selected to receive sanitation subsidy vouchers. Outcomes will be measured both for voucher recipients and for the rest of the community.

Inclusion Criteria (for Communities):

* Community was targeted by UNICEF's Community-Led Total Sanitation (CLTS) program in Tatale, Yendi, and Kpandai districts in Ghana.
* Community has Open Defecation Free (ODF) status according to local authorities.
* Community has more than 15 and less than 100 households.

Exclusion Criteria (for Communities):

* Community is located less than 2 kilometers away from a community in the opposite treatment arm.

Inclusion Criteria (for voucher recipients within study communities):

* Household is extremely poor, as identified through community consultation and/or the government's Livelihood Empowerment Against Poverty (LEAP) program.
* Household has at least one vulnerable person, i.e. who meets one of the following criteria: i) older than 65 years old, ii) person with a disability, iii) orphan or vulnerable child, iv) female head of household, v) widow(er), vi) terminally-ill persons, vii) unemployed, viii) outcast groups.

Exclusion Criteria (for voucher recipients within study communities):

* Household owns a functional, individual (non-shared) latrine with durable sub-structure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5615 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of households owning an individual, functional latrine with full superstructure | Approximately 18 months
  Household ownership (yes/no) of a latrine that is i) not shared with other households ("individual"), ii) whose pit is not collapsed and not full ("functional"), and iii) with four walls (or circular walls) and a roof of any materials ("full superstructure").

SECONDARY OUTCOMES:
Percentage of households reporting practicing open defecation | Approximately 18 months
  Self report by the respondent of not always using a toilet to defecate when at home.
Percentage of households owning an individual, functional latrine with full superstructure and durable superstructure | Approximately 18 months
  Household ownership (yes/no) of a latrine that is i) not shared with other households ("individual"), ii) whose pit is not collapsed and not full ("functional"), iii) with four walls (or circular walls) and a roof of any materials ("full superstructure"), iv) with a concrete/plastic slab and pit lining with plastic/rocks/bricks/concrete ("durable substructure").
Percentage of households reporting satisfaction with latrine | Approximately 18 months
  Self report by the respondent of being satisfied with the latrine (s)he uses for defecation.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Peletz, PhD, Principal Investigator — The Aquaya Institute
Locations (1):
- Districts of Tatale and Kpandai, Northern Region, Tamale, Ghana

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for the primary and all secondary outcome measures as well as key confounders (demographics, wealth index, community characteristics) will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 9 months of study completion.